CLINICAL TRIAL: NCT02717182
Title: Development of a Classification of the Components of Patient Therapeutic Education Interventions That Can Impact Their Results and Can Ensure Their Continued Existence CONCErTo Study
Brief Title: Classification of Patient Therapeutic Education Programs Components : Etude CONCErTo
Acronym: CONCErTo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: PREPS1439089
Record Dates: First submitted 2015-09-28; First posted 2016-03-23 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Chronic Disease
Keywords: self management program; patient education; self care program
MeSH Terms: conditions — Chronic Disease | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: interviews — interviews

SUMMARY:
Interest in patient therapeutic education (PTE) is increasing: in France PTE was included within the 2009 "Hospital, Patient, Health and Territory" law as an essential component of the patient healthcare pathway.

PTE is a complex intervention: its delivery is variable and may vary according to its content, functioning, providers, targeted patients, environment and even its objectives. These differences impact the expected results and make difficult the evaluation of PTE interventions. To overcome this difficulty, it is essential to describe precisely the intervention, the processes and the implementation of PTE that are usually not known. PTE interventions need today a global understanding of their mechanisms constituting their complexity.

CONCErTo study aims at developing a classification of the different elements composing a PTE intervention that can impact their results and can ensure their continued existence.

Mechanisms implemented during PTE interventions will be analyzed by a qualitative research. The investigators wish to identify organizational, pedagogical, psychosocial, medical or contextual elements that can impact the results, the patients' participation and the continuity of the program.

The perspective of this research is to improve the understanding of PTE by providing thorough description of the interventions. This work will help stakeholders to better interpret the results of their interventions, to improve the transferability, the implementation and finally to determine which are the elements able to improve patients' health status.

DETAILED DESCRIPTION:
This research is an observational study with no intervention. It uses qualitative methods.

The development of the classification consists in 3 phases: a preliminary phase of literature review, an investigation phase and a phase of elaboration of the classification.

Preliminary phase To deepen the questioning of the research, a literature review will be realized on concepts and models as well as on tools and methods used in the published PTE interventions.

Investigation phase

This step uses qualitative methods with 3 types of data collection:

* Semi structured interviews: individual interview will be realized with health care professionals and Therapeutic Patient Education stakeholders (trainers, professional network, decisions makers..). Focus groups will be organized with patients after completion of a therapeutic patient education program.
* In situ observations of the sessions
* Analysis of the documents surrounding the implementation of the interventions: reports, grey literature, applications; the objective is to capture the environment supervising the programs

The investigators plan to include up to 15 programs. However, this number will be adjusted according to the principle of data saturation.

Programs will be selected to ensure variability: the investigators will include hospital based or community based programs, programs led by general practitioners or specialists, with or without patients' implication, recent or experimented programs.

For each program, at least 3 health care professionals and one focus group with patients will be conducted. It will be completed by observation of education sessions.

Other actors (patients' proxies, associations playing a role in the conception or animation of the programs, designers, coordinators, general practitioners, experts of French territorial organization, trainers..;) will complete the data.

The aim of this step is not only to describe the practices but also to interview the experts on the elements they think can impact the results of PTE interventions.

Phase of elaboration of the classification Thematic and content data analyses are scheduled. Concept mapping method will be used to develop the classification.

The classification will be reviewed by experts having not participated to the previous steps.

Validation of the classification :

Applicability and relevance of the classification will be tested with 15 programs in various medical domains.

The classification will then be used in a cohort of patients before and after PTE intervention.

With this classification (or list), recommendations to describe PTE programs will be published.

Eventually, the aim of the recommendations, is to improve the understanding of PTE by providing thorough description of the interventions. This work will help stakeholders to better interpret the results of their interventions, to improve the transferability, the implementation and finally to determine which are the elements able to improve patients' health status.

ELIGIBILITY:
Inclusion Criteria:

* patients following a patient education program
* professionals involved in a patients education program

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients following a patient education program health care professionals
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Patient-reported elements of patient therapeutic education | 2 years
  Focus groups of patients
Heath care professionals-reported elements of patient therapeutic education | 2 years
  Individual Interviews of health care professionals

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Christine Rat, Principal Investigator — Nancy Hospital, CIC-EC Inserm CIC 1433; EA 4360 APEMAC
Locations (1):
- Rat Anne-Christine, Nancy, France